CLINICAL TRIAL: NCT01432340
Title: Seasonal Influenza Vaccine Effectiveness Study in the Kenyan Communities of Kibera and Lwak
Brief Title: Seasonal Influenza Vaccine Effectiveness Study in Kenya
Status: Completed | Type: Observational
Sponsor: Gideon Emukule (U.S. Federal Agency)
Collaborators: Kenya Ministry of Health (Other Government); Kenya Medical Research Institute (Other); Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Gideon Emukule, East Africa Influenza Program Director, Centers for Disease Control and Prevention
Organization: Centers for Disease Control and Prevention (U.S. Federal Agency)
Other Study IDs: CDC-NCIRD-5933
Record Dates: First submitted 2011-09-07; First posted 2011-09-12 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Influenza; Influenza Like Illness; Severe Acute Respiratory Illness
Keywords: Influenza; Influenza vaccine; Influenza vaccine effectiveness study
MeSH Terms: conditions — Influenza, Human | interventions — vaxigrip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal and oropharyngeal swabs.Potentially has DNA and RNA retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vaccinated group: Children between 6months- 10years of age who have received the influenza vaccine
  Interventions: Biological: Seasonal influenza vaccine
- Unvaccinated group: Eligible children between 6months and 10years who didn't receive the influenza vaccine
  Interventions: Biological: Seasonal influenza vaccine

INTERVENTIONS:
Biological: Seasonal influenza vaccine — annual recommended Southern Hemisphere vaccine
  Other Names: Vaxigrip

SUMMARY:
Influenza is an important cause of acute respiratory infections (ARI) worldwide. Seasonal influenza causes an estimated 250,000-500,000 deaths and 3-5 million severe illnesses each year (WHO, 2009), and pandemic 2009 H1N1 influenza has caused morbidity and mortality worldwide. In Kenya, influenza accounts for up to 50% of all ARI during the peak influenza season, based on Kenyan Ministry of Public Health and Sanitation and KEMRI/CDC surveillance data. Influenza vaccine has been shown to reduce influenza-associated ARIs in developed countries. However, little is know about the effectiveness of influenza vaccine in the developing world. In Kenya, a commercial trivalent injectable vaccine is licensed, but less than 30,000 doses are sold annually. The International Emerging Infections Program (IEIP) under KEMRI/CDC currently conducts population-based disease surveillance (PBDS) for severe acute respiratory illness (SARI) and influenza-like illness (ILI) in two sites in Kenya, Lwak (Nyanza province) and Kibera (Nairobi). The investigators propose to conduct a three-year influenza vaccine effectiveness study using the commercially available southern hemisphere seasonal vaccine for 2010, which includes the pandemic 2009 H1N1 component, and for 2011 and 2012. The study will evaluate the effectiveness of the vaccine in preventing laboratory-confirmed influenza, non-specific ARIs at the clinic and household level, and secondary influenza infection and secondary ARIs. Our study hypothesis is: Immunizing children with influenza vaccine will decrease influenza-associated acute respiratory infections among children and may reduce the number of non-specific acute respiratory infections in vaccinated children and their household contacts.

DETAILED DESCRIPTION:
Vaccine will be donated by Sanofi Pasteur in a quantity large enough to vaccinate the eligible population. Vaccine will be made available to infants from 6 months of age through children up to 10 years old. This includes an age group that is at high risk for severe outcomes (<5 years) and an age group (school-age children, 5-10) that is considered most likely to spread the infection.

Ascertainment of Influenza Illness:

Primary Outcome Measure

• Laboratory-confirmed influenza infection

Secondary outcome measures

* Medically attended ILI, SARI
* Community-reported ILI SARI
* Laboratory-confirmed influenza, medically attended ILI and SARI, and community-reported ILI and SARI in non-immunized household members

In Lwak and Kibera, field workers visit households weekly and encourage residents to go to the free clinic if they have respiratory symptoms. Currently, from KEMRI/CDC surveillance data, in Kibera, approximately 57 % of people in the catchment area seek medical care for ILI (Range: 62% children - 52% adults) and of those people who seek care, 72% seek care at Tabitha clinic. In Lwak, approximately 77% of people in the catchment area seek medical care for ILI (Range: 75% children - 80% adults) and of those people who seek care, 34% seek care at Lwak clinic.

The surveillance for ILI and SARI will continue as usual, with weekly field worker (also called community interviewer) household visits, clinic-based surveillance for ILI and SARI at Tabitha clinic and Lwak clinic, and sampling of all patients who meet the case definition for ILI and SARI

ELIGIBILITY:
Inclusion Criteria:

* Age 6months -10 years
* Enrolled in the IEIP morbidity study

Exclusion Criteria:

* Age less than 6 months or greater than or equal to 11 years
* Not enrolled in the IEIP morbidity study

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Vaccine will be made available to children six months of age to 10 years in the Kibera and Lwak catchment areas enrolled in the International Emerging Infectious Disease Program( IEIP) conducted by KEMRI/CDC.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2010-06; Primary Completion 2014-03-18 (Actual); Study Completion 2014-03-18 (Actual)

PRIMARY OUTCOMES:
Laboratory-confirmed influenza infection | June 2010-March 2013 (3 yrs)
  Look at the number of vaccinated children who develop laboratory-confirmed influenza infection compared to a matched unvaccinated group of children.

SECONDARY OUTCOMES:
Medically attended Influenza Like Illness(ILI) and Severe Acute Respiratory Illness (SARI) | June 2011-March 2013 (2 yrs)
  Look at the number of medically attended ILI and SARI in the unvaccinated group and compare to the vaccinated goup
Community-reported ILI SARI | June 2011- March 2013 (2 yrs)
  Look at the number of Community-reported ILI and SARI in the unvaccinated group and compare to the number in the vaccinated group
Laboratory-confirmed influenza, medically attended ILI and SARI, and community-reported ILI and SARI in non-immunized household members | June 2011-March 2013 (2 yrs)
  Look at the number of Laboratory-confirmed influenza, medically attended ILI and SARI, and community-reported ILI and SARI in non-immunized household members in both households that have a vaccinated child versus households that didn't have a vaccinated child

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Katz, MD, Principal Investigator — Center for Disease Control and Prevention-Kenya; Robert Breiman, MD, Principal Investigator — Centers for Disease Control and Prevention; Joshua Mott, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (2):
- Kenya (2):
  - KEMRI/CDC- IEIP surveillance-Asembo, Kisumu, Western
  - KEMRI/CDC IEIP surveillance- Kibera, Nairobi

REFERENCES:
- [Background] World Health Organization. Acute Respiratory Infections (Update September 2009). 2009. Available at http://www.who.int/vaccine_research/diseases/ari/en/print.html
- [Background] Williams BG, Gouws E, Boschi-Pinto C, Bryce J, Dye C. Estimates of world-wide distribution of child deaths from acute respiratory infections. Lancet Infect Dis. 2002 Jan;2(1):25-32. doi: 10.1016/s1473-3099(01)00170-0. PMID 11892493
- [Background] Viboud C, Alonso WJ, Simonsen L. Influenza in tropical regions. PLoS Med. 2006 Apr;3(4):e89. doi: 10.1371/journal.pmed.0030089. Epub 2006 Mar 7. PMID 16509764
- [Background] Belongia EA, Kieke BA, Donahue JG, Greenlee RT, Balish A, Foust A, Lindstrom S, Shay DK; Marshfield Influenza Study Group. Effectiveness of inactivated influenza vaccines varied substantially with antigenic match from the 2004-2005 season to the 2006-2007 season. J Infect Dis. 2009 Jan 15;199(2):159-67. doi: 10.1086/595861. PMID 19086915
- [Background] Center for Disease Control. ACIP Provisional Recommendations for the Use of Influenza Vaccines, March 2, 2010. Available at http://www.immunize.org/acip/